CLINICAL TRIAL: NCT07274891
Title: Comparative Evaluation of LigaSure Versus Bipolar Diathermy in Thyroidectomy: A Single-Center Study From Upper Egyp
Brief Title: LigaSure vs Bipolar Diathermy in Thyroidectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Keroles Atef Shaffik Nassem, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELVBDTSCSUE
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Thyroidectomy
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroidectomy using LigaSure (Active Comparator)
  Interventions: Procedure: LigaSure; Procedure: Thyroidectomy
- Thyroidectomy using bipolar diathermy (Active Comparator)
  Interventions: Procedure: bipolar diathermy; Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: LigaSure — LigaSure is an advanced vessel-sealing system that uses pressure and bipolar energy with real-time feedback to seal vessels up to 7 mm. It limits thermal spread, provides consistent sealing, and reduces the need for sutures-making it distinct from standard bipolar diathermy and other energy devices.
  Arms: Thyroidectomy using LigaSure
Procedure: bipolar diathermy — Bipolar diathermy uses two closely spaced electrodes to deliver controlled coagulation and cutting with minimal current spread. Unlike LigaSure or other advanced sealing devices, it lacks an automatic feedback system and does not fuse larger vessels, relying instead on direct thermal coagulation. It is simple, widely available, cost-effective, and suitable mainly for small-vessel hemostasis.
  Arms: Thyroidectomy using bipolar diathermy
Procedure: Thyroidectomy — Thyroidectomy is a standard surgical procedure for treating benign and malignant thyroid disorders.

SUMMARY:
Comparative Evaluation of LigaSure Versus Conventional Bipolar Diathermy in Thyroid Surgery: Operative and Postoperative Outcome.

DETAILED DESCRIPTION:
Thyroidectomy is a standard surgical procedure for treating benign and malignant thyroid disorders. Achieving precise hemostasis is essential to minimize intraoperative bleeding, preserve vital structures such as the recurrent laryngeal nerve and parathyroid glands, and prevent complications like hematoma and infection. Conventional bipolar diathermy has long been used to achieve hemostasis, but it can result in greater lateral thermal spread, prolonged operative time, and potential thermal injury to adjacent tissues.

LigaSure, an advanced vessel sealing system, combines pressure and energy to achieve permanent vessel fusion and can seal vessels up to 7 mm in diameter with minimal lateral thermal damage. Its use in thyroid surgery has been associated with improved surgical field visibility, reduced intraoperative bleeding, and shorter operative time compared to bipolar diathermy.

Additionally, LigaSure may lower the risk of postoperative complications, including transient hypocalcemia and recurrent laryngeal nerve palsy, due to its precise energy delivery and limited collateral damage.

However, existing studies have shown variable results regarding the magnitude of these benefits, and the cost-effectiveness of LigaSure compared with conventional bipolar diathermy remains uncertain. Therefore, a prospective randomized controlled trial is required to provide conclusive evidence regarding its role in reducing operative time and postoperative complications during thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) undergoing partial or total thyroidectomy.
2. Diagnosed with benign or low-risk malignant thyroid disorders.
3. Fit for general anesthesia.
4. Provided written informed consent to participate in the study.

Exclusion Criteria:

1.Previous neck surgery or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | during surgery 2 hours
  Total time (from skin to skin)Time taken for dissection and haemostasis
Number of ligatures used | during surgery

SECONDARY OUTCOMES:
Postoperative pain | 24 hours postoperative
  Pain assessment through the VAS was explained to the patient (through selection of the number that represents his/her pain with 0 = no pain, and 10 = worst pain
Transient or permanent hypocalcaemia | 24 hours postoperative

REFERENCES:
- [Result] Ali Alnnaser, Sulaiman J, Alloush A. A Comparative Study Between Total Thyroidectomy with Ligasure and Total Conventional Thyroidectomy. SRG International Journal of Medical Science. 2024 May;11(3):1-4
- [Result] Lee J, Nah KY, Kim RM, Ahn YH, Soh EY, Park CS. Comparison of the harmonic scalpel, LigaSure, and conventional technique in open thyroidectomy. Ann Surg Treat Res. 2016;90(2):61-66
- [Result] Markogiannakis H, Kekis PB, Memos N, Chatzimavroudis G, Lagoudianakis EE, Manouras A. Thyroid surgery using the electrothermal bipolar vessel sealing system. World J Surg. 2011;35(9):1962-1968
- [Result] Sakorafas GH, Stafyla V, Bramis K, Kotsifopoulos N, Kassaras GA. Ligasure versus clamp-and-tie thyroidectomy: a comparative study. Eur Surg Res. 2008;41(3):182-186
- [Result] Lachanas VA, Prokopakis EP, Mpenakis AA, Karatzanis AD, Velegrakis GA. LigaSure versus bipolar coagulation in total thyroidectomy. Am J Otolaryngol. 2014;35(6):766-770
- [Result] Kennedy JS, Stranahan PL, Taylor KD, Chandler JG. High-burst-strength, feedback-controlled bipolar vessel sealing. Surg Endosc. 1998 Jun;12(6):876-8. doi: 10.1007/s004649900733. PMID 9602010
- [Result] Dionigi G, Rovera F, Boni L, Castano P, Dionigi R. Electrothermal bipolar vessel sealing system (LigaSure) in thyroid surgery: a prospective, randomized study. Head Neck. 2010;32(6):718-722
- [Result] Yao HS, Wang Q, Wang WJ, Li J, Jin JW, Ma YY. A meta-analysis of LigaSure vs conventional vessel ligation in thyroidectomy. Surg Today. 2013;43(4):370-378